CLINICAL TRIAL: NCT02912663
Title: Magnesium And Verapamil After Recanalization in Ischemia of the Cerebrum (MAVARIC) in the Kentucky Regional Population: a Clinical and Translational Study.
Brief Title: Magnesium And Verapamil After Recanalization in Ischemia of the Cerebrum: a Clinical and Translational Study.
Acronym: MAVARIC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Justin Fraser (Other)
Responsible Party: Sponsor-Investigator, Justin Fraser, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Verapamil & magnisium sulfate
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Verapamil; Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Verapamil and Magnesium Sulfate (Experimental): 10mg of verapamil in 10 cc of normal saline and 1000mg of magnesium sulfate in 20cc of normal saline will be administered over 20 minutes (1cc/minute) through the microcatheter and into the vessel previously obstructed by clot to the treatment group
  Interventions: Drug: Verapamil and Magnesium Sulfate
- Placebo (Placebo Comparator): Control group will receive saline only
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Verapamil and Magnesium Sulfate — Single dose strategy will be used
  Arms: Verapamil and Magnesium Sulfate
Other: Placebo — Single matching dosing strategy will be used
  Other Names: 0.9% sodium chloride
  Arms: Placebo

SUMMARY:
This is a phase 1, blinded-outcome, randomized, placebo controlled study to investigate the safety and feasibility of super-selective intra-arterial administration of verapamil and magnesium sulfate immediately following successful endovascular thrombectomy as a potential neuroprotective synergistic therapeutic strategy in emergent large vessel occlusion stroke. This trial represents the first time that magnesium sulfate will be evaluated in human subjects as a superselectively administered neuroprotective agent administered in an acute time frame as an adjunct to intra-arterial thrombectomy. Furthermore, it will represent the first trial to evaluate combinational therapy for acute stroke neuroprotection.

DETAILED DESCRIPTION:
Participants will be recruited from patients evaluated at University of Kentucky Chandler Hospital for acute ischemic stroke. Participants with impaired capacity may be included, as the pathology to be studied (stroke) may impair their capacity. Initial contact will be made by the sub-investigators approved to obtain consent; all sub-investigators are practitioners who would make contact with potential participants in a clinical manner under standard clinical procedures. All sub-investigators will have access to stroke patients' medical information under normal circumstances. No special outreach is necessary to recruit particular populations. Enrollment goal will be 15 patients in each group.

Participants will not be compensated or provided any incentives for study participation.

The following describes all study procedures and evaluations that are to be done as part of the study.

Visit 1-Baseline (Day 0):

* Obtain consent.
* Medical history taken from medical record, participant and family to determine eligibility based on inclusion/exclusion criteria (Standard of Care)
* Medication history (Standard of Care)
* Physical examination to include vital signs (Standard of Care)
* Pregnancy Testing (Standard of Care)
* NIH Stroke Scale (Standard of Care)
* Verify inclusion/exclusion criteria
* Randomization
* Cerebral angiogram with Endovascular Thrombectomy (Standard of Care)
* Study Drug administration
* Adverse event (AE) collection

Immediately following the thrombectomy and study procedure all participants will be transferred to the Neuro-Intenstive care Unit (ICU) or other similar ICU for at least 24 hours for monitoring and care. Vital signs and neurological assessments will be assessed every hour. Evaluations of the groin access site will be performed every every 15 minutes for the first hour, then 30 minutes for the second hour, and finally every hour for the next 4 hours. Thereafter, groin site will be will performed at every shift.

Visit 2 - Within 48 hours of admission

• Non-contrast Postoperative MRI or CT (Standard of Care) The choice of one or the other will be determined by clinical criteria; CT or MRI may be preferable for different reasons depending upon the patient's clinical scenario.

Visit 3 - ( By Discharge)

* NIH Stroke Scale (Standard of Care)
* Discharge Destination (Standard of Care)
* Cognitive Assessment (Standard of Care)
* Radiographic assessment of primary and secondary radiologic endpoints

Visit 4 - End of Study (90 Days) (+/- 30 days)

* UBACC assessment will be used to assess consent capacity at follow-up.
* Montreal Cognitive Assessment (MoCA)
* Modified Rankin Score (mRS; Standard of Care)

The visit may be conducted over the phone with the participant or their legally authorized representative.

Unscheduled Visits. It is unexpected that Unscheduled Visits will be common, especially with the follow-up within 90 days after the procedure. However, subjects readmitted to the hospital for any reason will be tracked to determine if an AE occurred.

Prohibited Medications, Treatments and Procedures: Participants on therapeutic anticoagulation will be excluded from the study. If medically necessary for underlying conditions, therapeutic anticoagulation may be started 72 hours the study drug administration.

Participants should not use disopyramide within 48 hours before or 24 hours after verapamil and intravenous beta-block.

Following successful completion of the baseline visit, participants will be randomized into the study. The randomization number will be assigned by the PI/neurointerventionalist.

Participants will be randomized to receive 10mg of verapamil in 10 cc of normal saline and 1000mg of magnesium sulfate in 20cc of normal saline or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent and HIPAA form. Participants with impaired capacity may be included provided a Legally Authorized Representative as recognized by the the State of Kentucky, signs the informed consent.
* Willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged 18 years or older
* Suspected acute ischemic stroke based on clinical and radiographic evidence as determined and documented by the Stroke Neurology team at University of Kentucky.
* Participants must meet criteria for intra-arterial thrombectomy as determined and documented by Interventional Neuroradiology attending physician at University of Kentucky.
* Participants must have an acute thromboembolus within an intracranial artery in the anterior circulation (internal carotid, anterior cerebral, middle cerebral), which undergoes mechanical thrombectomy.
* Participant must have a TICI 2B or better revascularization via thrombectomy.
* For females of reproductive potential a negative pregnancy test at baseline is required.

Exclusion Criteria:

* Pregnant/lactating women
* Therapeutic anticoagulation prior to admission as it is a relative contraindication to thrombectomy
* Participants who undergo intra-arterial thrombectomy for acute stroke, in whom only TICI 0-2A revascularization is obtained.
* Known allergic reactions to components of Verapamil or magnesium sulfate.
* Verapamil should not be given to individuals who have a serious heart condition such as:

  * sick sinus syndrome or AV block
  * severe heart failure;
  * fainting do to slow heartbeats
  * certain heart rhythm disorders of the atrium (excluding atrial fibrillation)
  * active congestive heart failure;
  * low blood pressure;
  * a nerve-muscle disorder such as myasthenia gravis or muscular dystrophy.
* Magnesium Sulfate should not be given to individuals with heart block or heart damage.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-01-14 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Number of participants having no symptomatic intracranial hemorrhage | within 48 hours after treatment
  Defined as a hemorrhage occurring within 48 hours after study inclusion, temporally related to the intervention, and occurring with worsening neurological status as documented in the clinical exam.

SECONDARY OUTCOMES:
Number of participants who had no systemic side effects from verapamil and magnesium sulfate | within 90 days
  At any point during study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Justin Fraser, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Medical Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No